CLINICAL TRIAL: NCT05374707
Title: The Effect of Motivational Interviewing Technique on Smoking Urge and Smoking Cessation Success in Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ezgipasaoglu
Record Dates: First submitted 2022-04-23; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Smoking; Motivational Interviewing; School Health; Nursing
MeSH Terms: conditions — Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The sample of the study included the teachers working in six state secondary schools, which had the highest number of teachers among all secondary schools in Yunusemre and Şehzadeler districts and provided permission (n:446). Individuals who volunteered to participate in the study, did not have a malignant disease or a psychiatric problem, were non-smokers, and taught at schools included in the study were enrolled.
  The sample of the study consists of teachers working in six state secondary schools, which have the highest number of teachers among all secondary schools in the two central districts of a city and are allowed (n:446). Since schools were preferred as the randomization unit, three schools from six state secondary schools were determined as the experimental group and three schools as the control group by means of the random number generation software Research Randomizer.
Who Masked: Participant
Masking Description: He groups of smoking teachers were known by the researcher. In order to provide one sided blindness in the study, the smoking teachers were not informed about the groups to which their schools were assigned and therefore the groups they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The motivational interviewing group (Experimental): The data of the study were collected through online questionnaires. An motivational interviewing lasting 30 minutes on average, both online and face-to-face, was carried out with the experimental group. Four reminder text messages were sent to the experimental group in a one-month period.
  One month after the interview was carried out and Questionnaire on Smoking Urges and Smoking Cessation Success Prediction Scale were completed as a pretest for the experimental group, the scales were completed again as a post-test.
  Interventions: Behavioral: MOTIVATIONAL INTERVIEWING
- The group in which no motivational interviews were conducted (No Intervention): The control group, on the other hand, were asked to fill in Questionnaire on Smoking Urges and Smoking Cessation Success Prediction Scale as a pretest, and again a month later as a post-test.

INTERVENTIONS:
Behavioral: MOTIVATIONAL INTERVIEWING — Motivational interviewing is a form of interview conducted with a patient-centered approach in order to enable people to discover and solve the obstacles to behavior change.
  Arms: The motivational interviewing group

SUMMARY:
Background: Smoking, which remains one of the biggest public health threats that the world faces and has reached epidemic proportions, continues to cause more than eight million deaths on average per year worldwide. The aim of the study was to evaluate the effect of motivational interviewing technique on the smoking urge and the success of smoking cessation in teachers.

Methods: This was an experimental (randomized controlled) study where motivational interviews were conducted with the individuals in the experimental group. The sample of the study was chosen from the teachers, who met the inclusion criteria, in the secondary schools in the central districts of Manisa. The study was completed with 30 smokers in the experimental group and 31 smokers in the control group. Questionnaire on Smoking Urges, Smoking Cessation Success Prediction Scale and Sociodemographic Data Form were used as data collecting tools. Chi-square test, Mann-Whitney U test, Wilcoxon test, t-test and regression analysis were used to analyse the data.

ELIGIBILITY:
Criteria for inclusion

* Individuals who volunteered to participate in the study,
* Did not have a malignant disease or a psychiatric problem,
* Were smokers,
* Taught at schools included in the study were enrolled.

Exclusion criteria

* Those who did not volunteer to participate in the study
* Non-smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
The desire of individuals to smoke | 1 month
  Questionnaire on Smoking Urges: Measurement of smoking desires in experimental and control groups, before and after intervention. Scoring of the scale ranges from 10 to 70. The smallest score that can be obtained from the scale is 10, indicating no urge felt to quit smoking. The highest possible score is 70 and indicates a very high urge to smoke.
The achievements of individuals towards quitting smoking | 1 month
  Smoking Cessation Success Prediction Scale: Measurement of smoking cessation success before and after intervention in experimental and control groups. The lowest score that can be obtained from SCSPS is 10, and the highest is 50. Higher scores from the scale indicate higher success of smoking cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Mani̇sa, Turkey (Türkiye)